CLINICAL TRIAL: NCT06967506
Title: Assessment of the Blowing Exercises Using the Adjustable Personal Breathing Exercise Device AirOFit PRO™ in Children With Otitis Media With Effusion: A Randomized Prospective Controlled Trial
Brief Title: Evaluation of Blowing Exercises Utilizing a Breathing Exercise Device in Otitis Media With Effusion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44944914-2024
Record Dates: First submitted 2025-04-21; First posted 2025-05-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Otitis Media With Effusion (OME); Otitis Media With Effusion in Children; Breathing Exercise
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group with OME performing breathing exercises (Experimental): The blowing exercises to be performed with AirOFit PRO will be carried out as follows:
  1. Inhalation power will be adjusted: Using the device's own settings, inspiration will be performed with minimal effort for measurement. The participant will be asked to perform 3 maximum efforts at 30-second intervals, and the highest measured value will be recorded.
  2. Exhalation power: Using the device's own settings, expiration will be performed with maximum effort for measurement. The participant will be asked to perform 3 maximum efforts at 30-second intervals, and the highest measured value will be recorded.
  3. These exercises will be performed at least twice a day, preferably three times (morning/noon/evening).
  Interventions: Device: Blowing exercise group
- Control group (No Intervention): In this group, no blowing exercises will be performed apart from the routine OME treatment.

INTERVENTIONS:
Device: Blowing exercise group — Maximum effort exhalation exercises using the AirOFitPRO will be performed three times daily. Each session will be conducted for a minimum duration of five minutes, with 30-second intervals between each effort.
  Arms: The group with OME performing breathing exercises

SUMMARY:
Otitis media with effusion (OME) is a common condition in which fluid collects behind the eardrum without signs of infection. It can cause hearing problems and discomfort. Many children get better with medication, but in some cases, the condition becomes long-term and may require surgery.

OME is caused by dysfunction of the Eustachian tube, which helps balance the air pressure between the middle ear and the back of the nose (nasopharynx). Restoring proper airflow to the middle ear is important. In addition to medication, physicians often recommend pressure-based exercises such as balloon-blowing, swallowing exercises, the Valsalva maneuver, or chewing gum. These exercises help open the Eustachian tube by creating positive pressure in the nasopharynx, which can improve ear ventilation and reduce symptoms by relieving negative pressure in the middle ear.

This study will test the effect of a breathing exercise device called AirOFit PRO™ (AirOFit, Copenhagen, Denmark) in children with OME. Currently, there are no studies in the medical literature showing whether AirOFit PRO™ is effective in treating OME. If this study finds that using the AirOFit PRO™ helps children recover more quickly, it could be an important step in preventing chronic OME and reducing the need for surgery.

DETAILED DESCRIPTION:
Otitis media with effusion (OME) is one of the most common middle ear conditions in childhood. It is characterized by the presence of non-purulent fluid in the middle ear cavity without signs of acute infection. OME can cause conductive hearing loss, aural fullness, discomfort, and, in prolonged cases, delay in speech and language development. Many children improve with spontaneous resolution or standard medical therapy. However, some children develop chronic OME and may require surgical intervention such as tympanostomy tube insertion.

The main underlying mechanism in OME is Eustachian tube dysfunction. The Eustachian tube is responsible for pressure equalization and aeration of the middle ear. It opens physiologically during swallowing, yawning, and forceful nasal maneuvers. When Eustachian tube opening is insufficient, negative pressure develops in the middle ear and fluid may accumulate. Conservative management often includes behavioral or pressure-based exercises. These exercises include the Valsalva maneuver, balloon-blowing techniques, swallowing exercises, and chewing gum. The purpose of these maneuvers is to generate positive pressure in the nasopharynx. This positive pressure can facilitate Eustachian tube opening, improve middle ear ventilation, and help resolve effusion.

The AirOFit PRO™ (AirOFit, Copenhagen, Denmark) is a respiratory training device. It is designed to improve inhalation and exhalation performance by providing resistance-based breathing exercises. The device has mainly been used in sports and pulmonary rehabilitation contexts. There are no published clinical studies that investigate the effect of AirOFit PRO™ in children with OME. Since OME is closely related to impaired middle ear aeration, a device that delivers structured and measurable positive-pressure breathing exercises may have therapeutic potential in this population.

This randomized prospective controlled trial will evaluate the effectiveness of blowing exercises performed with the AirOFit PRO™ device in children aged 4 to 10 years with documented OME. Participants will be randomized into two groups. The intervention group will perform structured blowing exercises with AirOFit PRO™ in addition to routine OME management. The control group will receive routine OME treatment without any additional breathing or blowing exercises.

In the intervention group, inspiratory and expiratory resistance settings will first be adjusted using the device's own calibration procedure. Maximal inspiratory and expiratory efforts will be measured, and these values will guide the training settings. Participants will be instructed to perform maximum-effort expiratory exercises with the device at least twice daily and preferably three times daily. Sessions will be organized in the morning, at midday, and in the evening when feasible. Each session will last a minimum of five minutes. Efforts will be separated by standardized rest intervals of approximately 30 seconds between attempts.

The main objective of this study is to determine whether device-guided blowing exercises with AirOFit PRO™ shorten the time to resolution of OME compared with routine management alone. A positive result would support the use of this non-invasive, home-based intervention as an adjunctive treatment in children with OME. It could help reduce disease duration, lower the need for surgical procedures, and improve hearing-related quality of life in this age group. The findings may also contribute to future clinical practice guidelines on the conservative management of pediatric OME.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 10 years.
* Presence of documented OME findings in otoscopic examination and audiological measurements.
* Absence of any ear disease that could affect audiometric or tympanometric findings.
* Legal guardian consent must be obtained.

Exclusion Criteria:

* Presence of active upper respiratory infection symptoms.
* Presence of a chronic ear disease that could affect study outcomes (e.g., chronic otitis, tympanosclerosis, etc.).
* Presence of diseases affecting respiratory system functions (e.g., pneumonia, pleurisy, empyema, pneumothorax, hemothorax, hydrothorax, atelectasis, pulmonary edema, pulmonary hypertension, emphysema).
* Inability to perform respiratory exercises due to a general condition disturbance.
* Presence of psychomotor retardation that prevents the participant from performing blowing exercises.
* Refusal of the patient or their guardian to participate in the study without providing a reason.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Resolution of Tympanic Membrane Appearance and Normalization of Tympanometric Values | Participants will be followed weekly for up to 3 months after enrollment, or until resolution criteria are met, whichever occurs first.
  Participants' follow-up will be concluded upon achieving both (1) normalization of tympanic membrane appearance as determined by otoscopic examination (i.e., intact, translucent, and non-retracted membrane without signs of inflammation or effusion), and (2) tympanometric values within normal limits, defined as a Type A tympanogram [peak pressure between -100 and +50 decapascals (daPa), static acoustic compliance between 0.3 and 1.5 milliliters (mL), and external ear canal volume (ECV) within normal pediatric reference ranges for ages 4-10 years (0.3-1.0 mL)].

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak University Faculty of Medicine, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing personal data must comply with the data protection principles in Turkey.